# Document Cover Page

# Official Title of the Study:

Responsible Fatherhood Opportunities for Reentry & Mobility (ReFORM)

NCT Number: NCT02860988

**Date of Document:** September 29, 2020

Consent to Participate in a Research Study

#### **ReFORM PROGRAM EVALUATION**

January 2018

#### WHY ARE YOU BEING INVITED TO TAKE PART IN THIS RESEARCH?

You are being invited to take part in this study about understanding service needs among low-income, low-resource fathers who are involved in the criminal justice system. You are being invited to take part in this study because you are either 1) a participant in the MCCC sponsored workshops through the Administration of Children and Families (ACF), or, 2) an individual identified in a jail who has been identified as a father but the jails is not participating in the ACF supported workshops. If you volunteer to take part in this study, you will be one of about 650 men to do so over the next 5 years.

## WHO IS DOING THE STUDY?

The person in charge of the evaluation for this project is Matthew Webster, PhD of the University of Kentucky. There may be other people on the evaluation team assisting at different times during the study.

## WHAT IS THE PURPOSE OF THIS STUDY?

The purpose of this study is to examine the effectiveness of expanding Mountain Comprehensive Care (MCCC) services to improve employment options, father/child relationships, and overall well-being for individuals involved in the criminal justice system as they re-enter the community from jail.

## WHERE IS THE STUDY GOING TO TAKE PLACE AND HOW LONG WILL IT LAST?

The evaluation study will be conducted at one of three participating jail facilities including the Floyd County Detention Center (Prestonsburg), Big Sandy Regional Detention Center (Paintsville), and the Kentucky River Regional Detention Center (Hazard). During your incarceration, you will be asked to participate in 2 interviews. Follow-up interviews will also be conducted in the community post-release from jail (in-person, by telephone, or by Wi-Fi audio). Follow-up interviews in person will be conducted at public libraries, treatment facilities, and or offices at the University of Kentucky related 14 Community College libraries which are located throughout the state. You will need to come to one of these offices one time (6 months post-release) during the study for interviews. Each of those interviews will take about one hour. The total amount of time you will be asked to volunteer for this study is approximately three hours over the next year. If you are living in an institution (such as a treatment agency, hospital, jail, prison, etc.), study staff will attempt to conduct your follow-up interview at this facility.

## WHAT WILL YOU BE ASKED TO DO?

You will be asked to participate in an interview following your acceptance into the study based on your initial screening assessment. Your initial intake (and subsequent follow-up interviews) will include questions about employment history, family relationships, and income stability. In addition, your

interview will also include questions about factors which can influence those areas including drug and alcohol use, criminal behaviors, and mental health. You will be interviewed again at 3 months (or 12 weeks) post-intake and again 6 months post-release from jail in the community to answer similar types of questions. In addition to the locator information we collect at your first interview, the research team may also use other internet searches and social media sites like Facebook to try to find you for the follow-up. Your decision to enroll in any study related social media site is completely voluntary and your contact information will not be shared with any other study participant. Sites like Facebook (if you are a member) will just be used to send you notifications about your follow-up interview.

If you are involved in any services with MCCC during this study, you will also be asked for permission to include information from some of the clinical assessments that you complete at the program to be included in the evaluation. Each man who is invited to be a part of this evaluation study will receive the usual jail-supported services whether they volunteer to participate in the study or not. You may also be asked to take part in a voluntary focus group to provide information about your experiences in the areas of employment, income stability, and fatherhood.

## ARE THERE REASONS WHY YOU SHOULD NOT TAKE PART IN THIS STUDY?

There are no specific reasons that you would be excluded from voluntarily participating in this study.

# WHAT ARE THE POSSIBLE RISKS AND DISCOMFORTS?

Some of the interview questions that you will be asked are sensitive and personal, including drug and alcohol use, criminal activities, mental health, and family relationships. Talking about your past and present situations may make you feel uncomfortable. In addition, we may reveal information to the proper authorities if we believe you have abused a child, or you pose a danger to yourself, or to someone else. You do not have to answer any questions that you do not want to answer. You can stop answering questions or quit at any time and this will not affect your participation in services in any way. In addition to the risks listed above, you may experience a previously unknown risk or side effect.

## WILL YOU BENEFIT FROM TAKING PART IN THIS STUDY?

There is no guarantee that you will get any benefit from taking part in this study. However, your participation in this study may provide benefit to society by providing information related to treatment needs and treatment services for men who are reentering the community from jail. We cannot and do not guarantee that you will receive any benefit from taking part in this study.

## DO YOU HAVE TO TAKE PART IN THIS STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any benefits or rights you would normally have if you choose not to volunteer. You can stop at any time during the study and still keep the benefits and rights you had before volunteering. If you do not want to take part in this study, it won't affect your treatment status with any treatment/service agency or with any criminal justice agency, treatment, parole, or other agency. In addition, your decision to participate or not participate will in no way benefit or hurt your status with the prison system, Department of Corrections, or the parole board.

## IF YOU DON'T WANT TO TAKE PART IN THIS STUDY, ARE THERE OTHER CHOICES?

If you do not want to be in the study, there are no other choices except not to take part in the study. If you do not want to take part in this study, your participation in any treatment program or your probation/ parole status will not be affected.

## WHAT WILL IT COST YOU TO PARTICIPATE?

There is no charge to you for participating in the study.

## WHO WILL SEE THE INFORMATION THAT YOU GIVE?

Your information will be combined with information from other people taking part in the study. When we write about the study to share it with other researchers, we will write about the combined information we have gathered. You will not be identified in these write-ups. We may publish the results of this study; however, we will keep your name and other identifying information private. You will be asked for your social security number for payment of incentives.

We will make every effort to prevent anyone who is not on the evaluation team from knowing that you gave us information, or what that information is. For example, your name will be kept separate from the information you give, and these two things will be stored in different places under lock and key. You should know, however, that there are some circumstances in which we may have to show your information to other people. For example, we may reveal your information to the proper authorities if we believe you have abused a child, or you pose a danger to yourself or to someone else. In addition, someone at the Administration for Children and Families (ACF) and the University of Kentucky may look at or copy records that identify you. When results of this study are published, your name will not be used.

A Certificate of Confidentiality has been obtained from the US Department of Health and Human Services (DHHS) to protect the researchers from being forced, even by a court order or subpoena, to identify you. However, with the certificate, we may provide information to appropriate individuals or agencies if harm to you, harm to others, or child abuse or exploitation becomes a concern. The Certificate does not represent an endorsement of the research by the Secretary, DHHS. In addition, the agency funding this research (the Administration for Children and Families [ACF]), staff from the University of Kentucky and DHHS agencies may review records that identify you as part of their audit procedures.

Information that you provide in this study will not be shared with treatment providers or criminal justice officials. If you are currently on probation/parole, your participation in this study will not impact decisions made by your parole officers or other criminal justice authorities, and will not impact your parole status.

## CAN YOUR TAKING PART IN THE STUDY END EARLY?

If you decide to take part in the study, you still have the right to decide at any time that you no longer want to continue. No one will think badly of you or treat you differently if you decide not to take part in this study. The individuals conducting the study may need to withdraw you from the study. This may occur if you are not able to follow the directions they give you, if they find that your being in the study is

more risk than benefit to you, or if the agency funding the study decides to stop the study early for a variety of scientific reasons.

#### WILL YOU RECEIVE ANY REWARDS FOR TAKING PART IN THIS STUDY?

You will receive \$10 for taking part in the baseline interview and \$10 for each of follow-up interview at 3-months post intake and again at 6-months post-release from jail. If you are selected to participate and you agree to volunteer for the focus group, you will receive an additional \$10. Therefore, you have the opportunity to earn up to \$40 over the next year.

## WHAT IF YOU HAVE QUESTIONS?

Before you decide whether to take part in the study, please ask any questions that might come to mind now. Later, if you have questions about the study, you can contact the evaluator, Matthew Webster, Ph.D. (859-323-6100). If you have questions about your rights as a volunteer in this evaluation study, contact the staff in the Office of Research Integrity at the University of Kentucky at 859-257-9428 or toll free at 1-866-400-9428. We will give you a copy of this consent form to take with you.

The Administration for Children and Families (ACF) is providing financial support and/or material for this

## WHAT ELSE DO YOU NEED TO KNOW?

| study. You will be told if any new information is leaven willingness to continue taking part in this study | earned which may affect your condition or influence |
|---|---|
| Signature of person agreeing to take part in the stud | dy Date |
| Printed name of person taking part in the study | |
| Signature of person obtaining informed consent | Date |
| Signature of Investigator | |
| FOLLOW-UP PARTICIPATION You understand that you will be asked to participate and at 6 months post-release from jail as part of this responses will be strictly confidential, you understand you understand that participation is voluntary and y | s evaluation. You understand that all of your and that you will be paid for your participation, and |
| You agree to be contacted for follow-up interviews | for this evaluation. |
| Yes No | initials |

| FOLLOW-UP CONDI | TIONS | |
|---|---|---|
| You also understa | and that when the rese | earch assistant for this project attempts to contact you for a |
| follow-up intervie | ew, you may be living i | n another treatment facility, institution, prison, or jail. You |
| consent to being | contacted in any of the | ese facilities if the research assistant locates you for an interview. |
| _ | · | · · |
| Yes | No | initials |
| | <b></b> | |